CLINICAL TRIAL: NCT00139529
Title: Postpartum Maintenance of Abstinence From Tobacco
Brief Title: Education and Counseling for Abstinence From Tobacco After Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Patricia M. Risica, Asst Professor (Research), Brown University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 248; R01HL077608 (NIH)
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive an educational intervention during pregnancy combined with a motivational interviewing program using telephone counseling to prevent postpartum relapse to tobacco use.
  Interventions: Behavioral: Motivational Interviewing Telephone Counseling; Behavioral: Educational Intervention
- 2 (Active Comparator): Participants will receive an educational intervention during pregnancy.
  Interventions: Behavioral: Educational Intervention

INTERVENTIONS:
Behavioral: Motivational Interviewing Telephone Counseling — Participants will receive up to 5 phone calls.
  Arms: 1
Behavioral: Educational Intervention — Educational intervention will be completed during pregnancy.

SUMMARY:
The purpose of this study is to develop and field test a maintenance of smoking abstinence program designed for a predominately low-income, high-risk population of women from a wide variety of ethnic and racial backgrounds who have quit smoking because of (or during) their pregnancy.

DETAILED DESCRIPTION:
BACKGROUND:

Pregnancy is an ideal time to help underserved young women to stop smoking cigarettes and remain abstinent for life. The field has made great progress in assisting women to quit during this time. Unfortunately, maintenance of this highly significant behavior change is dismal. Up to 75% of those who quit for pregnancy end up returning to smoking after delivery of the newborn. For underserved women, pregnancy is one of the few times that they have an extended contact with the health care system. Therefore, there is an opportunity to help these women quit smoking for the health of their fetus in addition to their own health. To date, there has been insufficient research on how best to maintain abstinence during the critical postpartum period, during which a unique constellation of risk factors (including sleep deprivation, variations in negative mood, and increased stress) heighten the probability of relapse. The potential payoff is enormous. The literature, while not extensive, provides sufficient guidance and justification for the specific approach and intervention components the study has chosen.

DESIGN NARRATIVE:

This study will develop and field test a maintenance of smoking abstinence program to be designed for a predominately low-income, high-risk population of women from a wide variety of ethnic and racial backgrounds who have quit smoking because of (or during) their pregnancy. The study will compare biologically confirmed postpartum smoking relapse rates of women who receive an educational intervention during pregnancy combined with sustained telephone counseling after that intervention, with women who receive only an educational intervention. Participants will begin at 28 weeks prenatal and will be followed through 1, 3, 6, and 12 months postpartum.

The specific aims of the current maintenance study are: 1) to compare biochemically confirmed smoking abstinence rates of women who quit smoking during their pregnancy and who receive an intervention based on telephone counseling using motivational interviewing versus quitters who receive usual care, maintenance of abstinence will be assessed at 1, 3, 6, and 12 months postpartum; and 2) to collect both qualitative and quantitative data to better understand short term and long term maintenance mediators and moderators of abstinence postpartum for women of low socioeconomic status (SES) who quit smoking during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Smoked tobacco immediately before pregnancy

Exclusion Criteria:

* Smoked tobacco in the previous 7 days when contacted at 28 weeks gestation
* No telephone access

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 757 (Actual)
Dates: Start 2006-03; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Smoking status | Measured at 1, 3, 6, and 12 months postpartum
ETS exposure | Measured at 1, 3, 6, and 12 months postpartum
Urine cotinine analyses | Measured at 1, 3, 6, and 12 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M. Risica, DrPH, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States